CLINICAL TRIAL: NCT03272854
Title: TransplantLines Insulin Resistance and Inflammation Biobank and Cohort Study
Acronym: TxL-IRI
Status: Active, not recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Stephan J.L. Bakker, Internist-Neprologist, University Medical Center Groningen
Other Study IDs: METc2001/039
Record Dates: First submitted 2017-09-02; First posted 2017-09-06 (Actual); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Death; Graft Failure; Death, Cardiac; Diabetes
MeSH Terms: conditions — Death; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Biospecimen Retention: Samples Without DNA — EDTA plasma, serum, aliquots of 24h urine collections all stored at -80 degrees Centigrade.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Renal Transplant Recipients: A cohort or renal transplant recipients, all more than 1 year after transplantation at inclusion
  Interventions: Other: No intervention performed, the study is observational

INTERVENTIONS:
Other: No intervention performed, the study is observational

SUMMARY:
Short-term (1-year) results of renal transplantation are now excellent (over 95%). Long-term (10-year and longer) results are, however, still disappointing. Where most research has focused on immunosuppression and infections, the investigators hypothesize that in renal transplant recipient, amongst others overweight, obesity, chronic use of immunosuppressive drugs and impaired renal function contribute to insulin resistance and chronic low-grade inflammation, which pose the renal transplant recipients at increased risk for cardiovascular disease, decline of function of the transplanted kidney and other complications, including post-transplant diabetes. This study is a biobank and cohort study which investigates this hypothesis.

DETAILED DESCRIPTION:
Short-term (1-year) results of renal transplantation are now excellent (over 95%). Long-term (10-year and longer) results are, however, still disappointing. Where most research has focused on immunosuppression and infections, the investigators hypothesize that in renal transplant recipient, amongst others overweight, obesity, chronic use of immunosuppressive drugs and impaired renal function contribute to insulin resistance and chronic low-grade inflammation, which pose the renal transplant recipients at increased risk for cardiovascular disease, decline of function of the transplanted kidney and other complications, including post-transplant diabetes. To investigate this hypothesis we have detailedly phenotyped 606 renal transplant recipients who at the time of inclusion all were one year or more after transplantation, therewith providing a representation of stable outpatient renal trannsplant recipients late after renal transplantation. At the time of these baseline measurements, we also created a biobank with plasma, serum and aliquots of 24h urine collections. Beyond baseline, we have a regular update on adverse events, including all-cause mortality, cause-specific mortality, graft failure and development of new-onset diabetes after transplantation (NODAT).

ELIGIBILITY:
Inclusion Criteria:

* More than one year after renal transplantation
* History of renal transplantation

Exclusion Criteria:

* Signs of active infection
* Signs of active cardiac decompensation
* Active malignancy other than skin cancer
* Prognosis < 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stable outpatient renal transplant recipients more than 1 year after transplantation,
Sampling Method: Non-Probability Sample
Enrollment: 606 (Actual)
Dates: Start 2001-08 (Actual); Primary Completion 2003-07 (Actual); Study Completion 2031-08 (Estimated)

PRIMARY OUTCOMES:
All-Cause Mortality | 30 years
  All-Cause Mortality
Graft Failure | 30 years
  Death-Censored Graft Failure

SECONDARY OUTCOMES:
New Onset Diabetes After Transplantation | 30 years
  NODAT
Cardiovascular Mortality | 30 years
  Cause-Specific Mortality
Non-Cardiovascular Mortality | 30 years
  Cause-Specific Mortality

OTHER OUTCOMES:
Venous Thrombosis | 30 years
  Venous Thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Stephan JL Bakker, MD, PhD, Principal Investigator — University Medical Center Groningen

IPD SHARING:
Plan to Share IPD: Undecided
The data can be shared with other researchers. The researchers will then receive an anonymized dataset. The PI of the study will be co-author on papers that come out of the analyses.

REFERENCES:
- [Result] de Vries AP, Bakker SJ, van Son WJ, van der Heide JJ, Ploeg RJ, The HT, de Jong PE, Gans RO. Metabolic syndrome is associated with impaired long-term renal allograft function; not all component criteria contribute equally. Am J Transplant. 2004 Oct;4(10):1675-83. doi: 10.1111/j.1600-6143.2004.00558.x. PMID 15367224
- [Result] van Ree RM, de Vries AP, Oterdoom LH, The TH, Gansevoort RT, Homan van der Heide JJ, van Son WJ, Ploeg RJ, de Jong PE, Gans RO, Bakker SJ. Abdominal obesity and smoking are important determinants of C-reactive protein in renal transplant recipients. Nephrol Dial Transplant. 2005 Nov;20(11):2524-31. doi: 10.1093/ndt/gfi052. Epub 2005 Aug 22. PMID 16115856
- [Result] Oterdoom LH, de Vries AP, van Son WJ, van der Heide JJ, Ploeg RJ, Gansevoort RT, de Jong PE, Gans RO, Bakker SJ. Validation of insulin resistance indexes in a stable renal transplant population. Diabetes Care. 2005 Oct;28(10):2424-9. doi: 10.2337/diacare.28.10.2424. PMID 16186274
- [Result] Hartog JW, de Vries AP, Bakker SJ, Graaff R, van Son WJ, van der Heide JJ, Gans RO, Wolffenbuttel BH, de Jong PE, Smit AJ. Risk factors for chronic transplant dysfunction and cardiovascular disease are related to accumulation of advanced glycation end-products in renal transplant recipients. Nephrol Dial Transplant. 2006 Aug;21(8):2263-9. doi: 10.1093/ndt/gfl132. Epub 2006 Apr 5. PMID 16597636
- [Result] van Ree RM, Oterdoom LH, de Vries AP, Gansevoort RT, van der Heide JJ, van Son WJ, Ploeg RJ, de Jong PE, Gans RO, Bakker SJ. Elevated levels of C-reactive protein independently predict accelerated deterioration of graft function in renal transplant recipients. Nephrol Dial Transplant. 2007 Jan;22(1):246-53. doi: 10.1093/ndt/gfl511. Epub 2006 Sep 23. PMID 16998222
- [Result] Oterdoom LH, de Vries AP, Gansevoort RT, van Son WJ, van der Heide JJ, Ploeg RJ, de Jong PE, Gans RO, Bakker SJ. Determinants of insulin resistance in renal transplant recipients. Transplantation. 2007 Jan 15;83(1):29-35. doi: 10.1097/01.tp.0000245844.27683.48. PMID 17220787
- [Result] Oterdoom LH, de Vries AP, Gansevoort RT, de Jong PE, Gans RO, Bakker SJ. Fasting insulin modifies the relation between age and renal function. Nephrol Dial Transplant. 2007 Jun;22(6):1587-92. doi: 10.1093/ndt/gfm037. Epub 2007 Feb 21. PMID 17314207
- [Result] Gross S, van Ree RM, Oterdoom LH, de Vries AP, van Son WJ, de Jong PE, Navis GJ, Zuurman MW, Bierhaus A, Gans RO, Bakker SJ. Low levels of sRAGE are associated with increased risk for mortality in renal transplant recipients. Transplantation. 2007 Sep 15;84(5):659-63. doi: 10.1097/01.tp.0000280556.16275.2a. PMID 17876282
- [Result] van Timmeren MM, Vaidya VS, van Ree RM, Oterdoom LH, de Vries AP, Gans RO, van Goor H, Stegeman CA, Bonventre JV, Bakker SJ. High urinary excretion of kidney injury molecule-1 is an independent predictor of graft loss in renal transplant recipients. Transplantation. 2007 Dec 27;84(12):1625-30. doi: 10.1097/01.tp.0000295982.78039.ef. PMID 18165774
- [Result] Lijfering WM, de Vries AP, Veeger NJ, van Son WJ, Bakker SJ, van der Meer J. Possible contribution of cytomegalovirus infection to the high risk of (recurrent) venous thrombosis after renal transplantation. Thromb Haemost. 2008 Jan;99(1):127-32. doi: 10.1160/TH07-05-0340. PMID 18217144
- [Result] Oterdoom LH, van Ree RM, de Vries AP, Gansevoort RT, Schouten JP, van Son WJ, Homan van der Heide JJ, Navis G, de Jong PE, Gans RO, Bakker SJ. Urinary creatinine excretion reflecting muscle mass is a predictor of mortality and graft loss in renal transplant recipients. Transplantation. 2008 Aug 15;86(3):391-8. doi: 10.1097/TP.0b013e3181788aea. PMID 18698241
- [Result] van Ree RM, Oterdoom LH, de Vries AP, Homan van der Heide JJ, van Son WJ, Navis G, Gans RO, Bakker SJ. Circulating markers of endothelial dysfunction interact with proteinuria in predicting mortality in renal transplant recipients. Transplantation. 2008 Dec 27;86(12):1713-9. doi: 10.1097/TP.0b013e3181903d25. PMID 19104410
- [Result] Hartog JW, Gross S, Oterdoom LH, van Ree RM, de Vries AP, Smit AJ, Schouten JP, Nawroth PP, Gans RO, van Son WJ, Bierhaus A, Bakker SJ. Skin-autofluorescence is an independent predictor of graft loss in renal transplant recipients. Transplantation. 2009 Apr 15;87(7):1069-77. doi: 10.1097/TP.0b013e31819d3173. PMID 19352130
- [Result] Oterdoom LH, de Vries AP, van Ree RM, Gansevoort RT, van Son WJ, van der Heide JJ, Navis G, de Jong PE, Gans RO, Bakker SJ. N-terminal pro-B-type natriuretic peptide and mortality in renal transplant recipients versus the general population. Transplantation. 2009 May 27;87(10):1562-70. doi: 10.1097/TP.0b013e3181a4bb80. PMID 19461495
- [Result] van Ree RM, de Vries AP, Oterdoom LH, Seelen MA, Gansevoort RT, Schouten JP, Struck J, Navis G, Gans RO, van der Heide JJ, van Son WJ, Bakker SJ. Plasma procalcitonin is an independent predictor of graft failure late after renal transplantation. Transplantation. 2009 Jul 27;88(2):279-87. doi: 10.1097/TP.0b013e3181ac9ea0. PMID 19623026
- [Result] van Ree RM, de Vries AP, Zelle DM, de Vries LV, Oterdoom LH, Gans RO, Schouten JP, Lems SP, van Son WJ, Bakker SJ. Latent cytomegalovirus infection is an independent risk factor for late graft failure in renal transplant recipients. Med Sci Monit. 2011 Nov;17(11):CR609-617. doi: 10.12659/msm.882045. PMID 22037739
- [Result] Said MY, Deetman PE, de Vries AP, Zelle DM, Gans RO, Navis G, Joosten MM, Bakker SJ. Causal path analyses of the association of protein intake with risk of mortality and graft failure in renal transplant recipients. Clin Transplant. 2015 May;29(5):447-57. doi: 10.1111/ctr.12536. Epub 2015 Apr 23. PMID 25739949
- [Result] Eisenga MF, Dullaart RP, Berger SP, Sloan JH, de Vries AP, Bakker SJ, Gaillard CA. Association of hepcidin-25 with survival after kidney transplantation. Eur J Clin Invest. 2016 Dec;46(12):994-1001. doi: 10.1111/eci.12682. Epub 2016 Oct 26. PMID 27696386
- [Result] Adepu S, Katta K, Tietge UJ, Kwakernaak AJ, Dam W, van Goor H, Dullaart RP, Navis GJ, Bakker SJ, van den Born J. Hepatic syndecan-1 changes associate with dyslipidemia after renal transplantation. Am J Transplant. 2014 Oct;14(10):2328-38. doi: 10.1111/ajt.12842. Epub 2014 Aug 25. PMID 25154787
- [Result] Annema W, Dikkers A, de Boer JF, Dullaart RP, Sanders JS, Bakker SJ, Tietge UJ. HDL Cholesterol Efflux Predicts Graft Failure in Renal Transplant Recipients. J Am Soc Nephrol. 2016 Feb;27(2):595-603. doi: 10.1681/ASN.2014090857. Epub 2015 Aug 28. PMID 26319244
- [Result] Leberkuhne LJ, Ebtehaj S, Dimova LG, Dikkers A, Dullaart RP, Bakker SJ, Tietge UJ. The predictive value of the antioxidative function of HDL for cardiovascular disease and graft failure in renal transplant recipients. Atherosclerosis. 2016 Jun;249:181-5. doi: 10.1016/j.atherosclerosis.2016.04.008. Epub 2016 Apr 8. PMID 27107804
- [Result] Eisenga MF, Zelle DM, Sloan JH, Gaillard CAJM, Bakker SJL, Dullaart RPF. High Serum PCSK9 Is Associated With Increased Risk of New-Onset Diabetes After Transplantation in Renal Transplant Recipients. Diabetes Care. 2017 Jul;40(7):894-901. doi: 10.2337/dc16-2258. Epub 2017 May 1. PMID 28461454
- [Result] Eisenga MF, Dullaart RPF, Berger SP, Touw DJ, Bakker SJL, Gaillard CAJM. Urinary prednisolone excretion is a determinant of serum hepcidin levels in renal transplant recipients. Am J Hematol. 2017 Aug;92(8):E173-E175. doi: 10.1002/ajh.24785. Epub 2017 Jun 9. No abstract available. PMID 28494514
- [Result] Sotomayor CG, Eisenga MF, Gomes Neto AW, Ozyilmaz A, Gans ROB, Jong WHA, Zelle DM, Berger SP, Gaillard CAJM, Navis GJ, Bakker SJ. Vitamin C Depletion and All-Cause Mortality in Renal Transplant Recipients. Nutrients. 2017 Jun 2;9(6):568. doi: 10.3390/nu9060568. PMID 28574431
- [Result] van Timmeren MM, Lems SP, Hepkema BG, Bakker SJ. Anti-human leukocyte antigen antibodies and development of graft failure after renal transplantation. Transplantation. 2009 Dec 27;88(12):1399-400. doi: 10.1097/TP.0b013e3181bc3ef0. No abstract available. PMID 20029338
- [Result] Zelle DM, Corpeleijn E, van Ree RM, Stolk RP, van der Veer E, Gans RO, Homan van der Heide JJ, Navis G, Bakker SJ. Markers of the hepatic component of the metabolic syndrome as predictors of mortality in renal transplant recipients. Am J Transplant. 2010 Jan;10(1):106-14. doi: 10.1111/j.1600-6143.2009.02876.x. Epub 2009 Nov 24. PMID 19951280
- [Result] van Ree RM, Gross S, Zelle DM, van der Heide JJ, Schouten JP, van Son WJ, Gans RO, Bakker SJ. Influence of C-reactive protein and urinary protein excretion on prediction of graft failure and mortality by serum albumin in renal transplant recipients. Transplantation. 2010 May 27;89(10):1247-54. doi: 10.1097/TP.0b013e3181d720e3. PMID 20559032
- [Result] Zelle DM, Corpeleijn E, Stolk RP, de Greef MH, Gans RO, van der Heide JJ, Navis G, Bakker SJ. Low physical activity and risk of cardiovascular and all-cause mortality in renal transplant recipients. Clin J Am Soc Nephrol. 2011 Apr;6(4):898-905. doi: 10.2215/CJN.03340410. Epub 2011 Mar 3. PMID 21372213
- [Result] Agarwal PK, Hellemons ME, Zelle DM, van Ree RM, van den Born J, van der Heide JJ, Gans RO, van Son WJ, Navis G, Bakker SJ. Smoking is a risk factor for graft failure and mortality after renal transplantation. Am J Nephrol. 2011;34(1):26-31. doi: 10.1159/000328903. Epub 2011 Jun 9. PMID 21659736
- [Result] Zelle DM, Agarwal PK, Ramirez JL, van der Heide JJ, Corpeleijn E, Gans RO, Navis G, Bakker SJ. Alcohol consumption, new onset of diabetes after transplantation, and all-cause mortality in renal transplant recipients. Transplantation. 2011 Jul 27;92(2):203-9. doi: 10.1097/TP.0b013e318222ca10. PMID 21685828
- [Result] Sinkeler SJ, Zelle DM, Homan van der Heide JJ, Gans RO, Navis G, Bakker SJ. Endogenous plasma erythropoietin, cardiovascular mortality and all-cause mortality in renal transplant recipients. Am J Transplant. 2012 Feb;12(2):485-91. doi: 10.1111/j.1600-6143.2011.03825.x. Epub 2011 Nov 4. PMID 22054202
- [Result] Deetman PE, Zelle DM, Homan van der Heide JJ, Navis GJ, Gans RO, Bakker SJ. Plasma bilirubin and late graft failure in renal transplant recipients. Transpl Int. 2012 Aug;25(8):876-81. doi: 10.1111/j.1432-2277.2012.01515.x. Epub 2012 Jun 21. PMID 22716194
- [Result] Zelle DM, Dorland HF, Rosmalen JG, Corpeleijn E, Gans RO, Homan van der Heide JJ, van Son WJ, Navis G, Bakker SJ. Impact of depression on long-term outcome after renal transplantation: a prospective cohort study. Transplantation. 2012 Nov 27;94(10):1033-40. doi: 10.1097/TP.0b013e31826bc3c8. PMID 23064656
- [Result] Zelle DM, Corpeleijn E, Deinum J, Stolk RP, Gans RO, Navis G, Bakker SJ. Pancreatic beta-cell dysfunction and risk of new-onset diabetes after kidney transplantation. Diabetes Care. 2013 Jul;36(7):1926-32. doi: 10.2337/dc12-1894. Epub 2013 Feb 1. PMID 23378624
- [Result] Zelle DM, Corpeleijn E, Klaassen G, Schutte E, Navis G, Bakker SJ. Fear of Movement and Low Self-Efficacy Are Important Barriers in Physical Activity after Renal Transplantation. PLoS One. 2016 Feb 4;11(2):e0147609. doi: 10.1371/journal.pone.0147609. eCollection 2016. PMID 26844883
- [Result] Hellemons ME, Sanders JS, Seelen MA, Gans RO, Muller Kobold AC, van Son WJ, Postmus D, Navis GJ, Bakker SJ. Assessment of Cotinine Reveals a Dose-Dependent Effect of Smoking Exposure on Long-term Outcomes After Renal Transplantation. Transplantation. 2015 Sep;99(9):1926-32. doi: 10.1097/TP.0000000000000636. PMID 25710609
- [Result] Meijer E, Bakker SJ, de Jong PE, Homan van der Heide JJ, van Son WJ, Struck J, Lems SP, Gansevoort RT. Copeptin, a surrogate marker of vasopressin, is associated with accelerated renal function decline in renal transplant recipients. Transplantation. 2009 Aug 27;88(4):561-7. doi: 10.1097/TP.0b013e3181b11ae4. PMID 19696640
- [Result] Nauta FL, Bakker SJ, van Oeveren W, Navis G, van der Heide JJ, van Goor H, de Jong PE, Gansevoort RT. Albuminuria, proteinuria, and novel urine biomarkers as predictors of long-term allograft outcomes in kidney transplant recipients. Am J Kidney Dis. 2011 May;57(5):733-43. doi: 10.1053/j.ajkd.2010.12.022. Epub 2011 Apr 1. PMID 21458900
- [Result] de Vries LV, Minovic I, Franssen CFM, van Faassen M, Sanders JS, Berger SP, Navis G, Kema IP, Bakker SJL. The tryptophan/kynurenine pathway, systemic inflammation, and long-term outcome after kidney transplantation. Am J Physiol Renal Physiol. 2017 Aug 1;313(2):F475-F486. doi: 10.1152/ajprenal.00690.2016. Epub 2017 May 10. PMID 28490533
- [Result] Keyzer CA, Riphagen IJ, Joosten MM, Navis G, Muller Kobold AC, Kema IP, Bakker SJ, de Borst MH; NIGRAM consortium. Associations of 25(OH) and 1,25(OH)2 vitamin D with long-term outcomes in stable renal transplant recipients. J Clin Endocrinol Metab. 2015 Jan;100(1):81-9. doi: 10.1210/jc.2014-3012. PMID 25361179
- [Result] Keyzer CA, Vermeer C, Joosten MM, Knapen MH, Drummen NE, Navis G, Bakker SJ, de Borst MH. Vitamin K status and mortality after kidney transplantation: a cohort study. Am J Kidney Dis. 2015 Mar;65(3):474-83. doi: 10.1053/j.ajkd.2014.09.014. Epub 2014 Nov 12. PMID 25453995
- [Result] Baia LC, Humalda JK, Vervloet MG, Navis G, Bakker SJ, de Borst MH; NIGRAM Consortium. Fibroblast growth factor 23 and cardiovascular mortality after kidney transplantation. Clin J Am Soc Nephrol. 2013 Nov;8(11):1968-78. doi: 10.2215/CJN.01880213. Epub 2013 Aug 8. PMID 23929933
- [Derived] Anderson JLC, Bakker SJL, Tietge UJF. The triglyceride to HDL-cholesterol ratio and chronic graft failure in renal transplantation. J Clin Lipidol. 2021 Mar-Apr;15(2):301-310. doi: 10.1016/j.jacl.2021.01.009. Epub 2021 Feb 2. PMID 33589404
- [Derived] Sotomayor CG, Te Velde-Keyzer CA, Diepstra A, van Londen M, Pol RA, Post A, Gans ROB, Nolte IM, Slart RHJA, de Borst MH, Berger SP, Rodrigo R, Navis GJ, de Boer RA, Bakker SJL. Galectin-3 and Risk of Late Graft Failure in Kidney Transplant Recipients: A 10-year Prospective Cohort Study. Transplantation. 2021 May 1;105(5):1106-1115. doi: 10.1097/TP.0000000000003359. PMID 32639409
- [Derived] Szili-Torok T, Bakker SJL, Tietge UJF. Statin Use Is Prospectively Associated With New-Onset Diabetes After Transplantation in Renal Transplant Recipients. Diabetes Care. 2020 Aug;43(8):1945-1947. doi: 10.2337/dc19-1212. Epub 2020 May 22. PMID 32444455
- [Derived] Sotomayor CG, Gomes-Neto AW, van Londen M, Gans ROB, Nolte IM, Berger SP, Navis GJ, Rodrigo R, Leuvenink HGD, Schalkwijk CG, Bakker SJL. Circulating Advanced Glycation Endproducts and Long-Term Risk of Cardiovascular Mortality in Kidney Transplant Recipients. Clin J Am Soc Nephrol. 2019 Oct 7;14(10):1512-1520. doi: 10.2215/CJN.00540119. Epub 2019 Sep 17. PMID 31530552
- [Derived] Szili-Torok T, Annema W, Anderson JLC, Bakker SJL, Tietge UJF. HDL Cholesterol Efflux Predicts Incident New-Onset Diabetes After Transplantation (NODAT) in Renal Transplant Recipients Independent of HDL Cholesterol Levels. Diabetes. 2019 Oct;68(10):1915-1923. doi: 10.2337/db18-1267. Epub 2019 Aug 2. PMID 31375510
- [Derived] Sotomayor CG, Gomes-Neto AW, Eisenga MF, Nolte IM, Anderson JLC, de Borst MH, Oste MCJ, Rodrigo R, Gans ROB, Berger SP, Navis GJ, Bakker SJL. Consumption of fruits and vegetables and cardiovascular mortality in renal transplant recipients: a prospective cohort study. Nephrol Dial Transplant. 2020 Feb 1;35(2):357-365. doi: 10.1093/ndt/gfy248. PMID 30165500